CLINICAL TRIAL: NCT03961503
Title: Acute Kidney Injury During Daptomycin Versus Vancomycin Treatment in Cardiovascular Critically Ill Patients: a Propensity Score Matched Analysis
Brief Title: Retrospective Analysis of Nephrotoxicity During Daptomycin Versus Vancomycin Treatments in High Risk Patients
Acronym: DVN
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: Q-2015-05-03
Record Dates: First submitted 2019-05-16; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Infective Endocarditis; Infection Related to Ventricular Assist Device; Infection Related to Vascular Prothesis; Surgical Site Infection; Mediastinitis
Keywords: Vancomycin; Daptomycin; Acute Kidney Injury; Nephrotoxicity; Infective Endocarditis; Foreign Body Associated Infection; Cardiovascular surgery
MeSH Terms: conditions — Endocarditis; Surgical Wound Infection; Mediastinitis; Acute Kidney Injury | interventions — Daptomycin; Therapeutics; Vancomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Plasma: preoperative, ICU admission at POD0 and POD1 samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Daptomycin (DAP): DAP : Cohort of patients who received daptomycin as the first line treatment for at least 48 hours for the defined indication
  Interventions: Drug: Daptomycin (DAP) treatment
- Vancomycin (VAN): VAN : Cohort of patients who received vancomycin as the first line treatment for at least 48 hours for the defined indication
  Interventions: Drug: Vancomycin (VAN) treatment

INTERVENTIONS:
Drug: Daptomycin (DAP) treatment — Group DAP : Daptomycin was administered at a dose of 8 mg/kg in thirty-minutes intravenous infusion every 24 hours in patients without severe impairment of kidney function or every 48 hours in case of GFR below 30 ml/min/m2. The creatine-kinase (CK) level was measured before the initiation of DAP and at least once a week to assess the occurrence of muscular toxicity defined by an increase of CK up to 3-fold the upper superior limit without any evidence of member ischaemia.
  Other Names: Group DAP
  Groups: Daptomycin (DAP)
Drug: Vancomycin (VAN) treatment — Group VAN : Vancomycin intravenous treatment was initiated by a loading dose of 30 mg/kg in 1 hour and followed by a continuous maintenance infusion dosing between 15 and 30 mg/kg/d. The VAN dose was adapted to achieve a target serum vancomycin steady-state concentration of 20-30 mg/L assessed by a daily pharmacologic monitoring (therapeutic drug monitoring).
  Other Names: Group VAN
  Groups: Vancomycin (VAN)

SUMMARY:
Acute kidney injury (AKI) is a frequent complication that occurs in 15 to 25% of patients after vascular surgery, and up to 40% of patients after cardiac surgery. AKI compromises seriously short and long-term prognosis of critically ill patients. Several AKI risk factors have been identified including a chronic pathology of the patient such as kidney failure or diabetes, acute kidney injury related to hemodynamic disorders during surgery, including cardiopulmonary bypass, or sepsis, and the use of nephrotoxic agents such as some antibiotics, colloids or iodine contrast agents. Avoiding nephrotoxic agents is therefore strongly recommended in ICU patients, to reduce the incidence of AKI, or to reduce its severity.

The aim of this cohort study was to assess whether the use of daptomycin, was associated to a lower incidence of AKI than vancomycin in cardiovascular ICU patients, with similar efficacy.

This is a retrospective observational study with a propensity score adjustment to reduce the bias of selection for a comparative analysis between two antibacterial treatments used in routine care.

Since treatments were not randomized, the investigators used the propensity score method for primary endpoint analysis. For this, the investigators included the covariates potentially related to treatment and outcome in a multivariate logistic model explaining the choice of treatment. This propensity score was used in the second model as an adjustment covariate included in the multivariate analysis to determine factors independently associated with the primary endpoint (AKI within 7 days).

The main hypothesis is the first line antibiotic treatment with daptomycin leads to less nephrotoxicity than vancomycin in a population known at high risk for AKI and with at least a similar efficacy on clinical success rate.

ELIGIBILITY:
Inclusion criteria:

* Patient older than 18 years
* Admitted in ICU from January 2010 to December 2012
* Suspected or proven cardiac, vascular or profound surgical site infection with Gram-positive cocci (GPC) methicillin-resistant (MR) strains (including probabilistic treatment for patients with acquisition of MR risk factors)
* Treatment duration greater than or equal to 48 hours (at least 2 doses of daptomycin administered or 2 days of vancomycin infusion)
* Antibiotic treatment started in peri-operative (from 48 hours before the onset of surgery) or in postoperative period (during ICU stay)

Exclusion criteria:

* Prophylaxis indication of antibiotics
* Kidney disease on chronic dialysis
* Acute onset of RRT before initiation of DAP or VAN treatment
* Staphylococcus pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted in Intensive Care Unit before and/or after cardiovascular surgery with at least one organ failure
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-01-30 (Actual); Study Completion 2016-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Acute Kidney Injury (AKI) | 7 days after the treatment initiation
  AKI stade 1, 2 or 3 according to KDIGO definition with baseline creatinine given by the last creatinine value before the start of treatment

SECONDARY OUTCOMES:
Incidence of Acute Kidney Injury (AKI) | 14 days after the treatment initiation
  AKI stade 1, 2 or 3 according to KDIGO definition with baseline creatinine given by the last creatinine value before the start of treatment
Maximal decrease of glomerular filtration rate (GFR) | Through study treatment completion, an average of 2 weeks
  Decrease of GFR, estimated by CKD-EPI formula, from baseline as measured by all serum creatinine determinations during treatment
Incidence of severe renal failure | Through study treatment completion, an average of 2 weeks
  AKI stade 2 or 3 according to KDIGO definition or decrease of GFR more than 50% from baseline
Incidence of renal replacement therapy (RRT) | Through study treatment completion, an average of 2 weeks
  RRT initiated between the first and the last treatment administrations
Duration of RRT | Through study completion limited to ICU stay, an average of 2 weeks
  Number of days between the first RRT initiation and the end of the last RRT during the ICU stay (excluding RRT performed in a dialysis center for chronic renal failure)
Incidence of clinical treatment failure | 15 days after the end of treatment
  defined by either persistent positive cultures, worsening of clinical status, death due to initial infection, or relapse after the end of treatment. It was assessed in case of documented GPC infection
Incidence of premature discontinuation of treatment | Through study treatment completion, an average of 2 weeks
  defined as a treatment stopped because of adverse event or clinical failure except death
Mortality | 28 days after treatment initiation
  all cause mortality
Mortality | 6 months (180 days) after treatment initiation
  all cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gaudard, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No